CLINICAL TRIAL: NCT07234396
Title: Animated Procedure Video Reduces Pain and Anxiety Among Pediatric Patients Undergoing Pin Removal Following Supracondylar Fracture Fixation - A Randomized Controlled Trial
Brief Title: Animated Video and Associated Pain and Anxiety Reduction, Following Pin Removal Post-supracondylar Fracture Fixation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat National Hospital & Medical College (Other)
Responsible Party: Principal Investigator, Mohammad Zeeshan Haider, Resident Doctor, Liaquat National Hospital & Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: RC-LNH-Orthopedics-10/2025/126
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Supracondylar Fractures; Fracture Fixation; Pain Severity; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients undergoing pin removal being shown an animated video of the procedure. (Experimental): Patients undergoing K-wire removal after fixation of supracondylar fractures being shown an animated video of the procedure while it is performed.
  Interventions: Procedure: K-wire removal with animated procedure video being shown to the patient during its performance.
- Patients undergoing pin removal without being shown an animated video of the procedure. (Active Comparator): Patients undergoing K-wire removal after fixation of supracondylar fractures without being shown an animated video of the procedure while it is performed.
  Interventions: Procedure: K-wire removal without animated procedure video being shown to the patient during its performance.

INTERVENTIONS:
Procedure: K-wire removal with animated procedure video being shown to the patient during its performance. — K-wire removal, post-supracondylar fracture fixation, will be performed while showing the patient an animated video of the procedure.
  Arms: Patients undergoing pin removal being shown an animated video of the procedure.
Procedure: K-wire removal without animated procedure video being shown to the patient during its performance. — K-wire removal, post-supracondylar fracture fixation, will be performed without showing the patient an animated video of the procedure.
  Arms: Patients undergoing pin removal without being shown an animated video of the procedure.

SUMMARY:
Assessing the reduction in pain and anxiety by the use of showing an animated video of the procedure, among pediatric patients undergoing pin removal after fixation of supracondylar fractures.

DETAILED DESCRIPTION:
Supracondylar fractures requiring K-wire fixation ultimately undergo pin removal after fracture fixation. This is a cause of pain and anxiety to children. This study aims to curtail the aforementioned troubles by distracting the patient using an animated video of the procedure. Patients will be randomized into two arms, and pain and anxiety scales will be implemented before, during, and after the procedure to assess whether a change exists between the two arms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with supracondylar fractures operated on for percutaneous K-wire fixation.
* Age between 4 to 12 years

Exclusion Criteria:

* Any syndromic patients
* Patients having any visual or cognitive disability
* Patients having any pre-operative or post-operative complications before pin removal.
* Patients undergoing the procedure under general anesthesia.
* Age <4 or >12

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Wong Baker Pain scale (WBS) | Evaluation will be done as per the criteria before, during the standard procedure, and 60 minutes post-procedure.
  The Wong Baker Pain scale will be used to assess pain before, during, and after the procedure being performed. A self-assessment tool for pain that uses six cartoon faces to grade pain on a numerical range of 0-10 ranked in increasing order of pain. Higher scores depict worse outcome and increased pain.
Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) | Evaluation will be done as per the criteria before, during the standard procedure, and 60 minutes post-procedure.
  Children's Hospital of Eastern Ontario Pain Scale will be used to assess pain before, during, and after the procedure being performed. A 10-item observational tool used to assess postoperative pain from a score of 4 to 13, higher scores indicating more pain and worse outcome.
Children's Anxiety Meter-State (CAM-S) | Evaluation will be done as per the criteria before, during the standard procedure, and 60 minutes post-procedure.
  The Children's Anxiety Meter-State scale will be used to assess anxiety before, during, and after the procedure being performed. This is a brief measure where scores are on a scale of 0-10; low scores depict better outcomes and high scores depict worse outcomes.
Short State Trait Anxiety Inventory Scale (STAI) | Evaluation will be done as per the criteria before, during the standard procedure, and 60 minutes post-procedure.
  The Short State Inventory Scale will be used to assess anxiety before, during, and after the procedure being performed, using the questionnaire set by the scale itself. A 20-item self reported assessment tool which scores each item from 1 to 4 for a minimum score of 20 to a maximum of 80. Low scores mean less anxiety and better outcome and a high score means greater anxiety and worse outcome. Positively phrased items are reverse-scored to calculate the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Nabeel Aamir Syed, MBBS, MD, Principal Investigator
Locations (1):
- Liaquat National Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No